CLINICAL TRIAL: NCT01109693
Title: Strategic Use of New Generation Antidepressants for Depression
Acronym: SUN(^_^)D
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyoto University (Other)
Collaborators: National Center of Neurology and Psychiatry, Japan (Other)
Responsible Party: Principal Investigator, Toshiaki A. Furukawa, Professor, Kyoto University
Organization: Kyoto University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sun-d
Record Dates: First submitted 2010-04-21; First posted 2010-04-23 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Unipolar Major Depressive Episode
MeSH Terms: interventions — Sertraline; Mirtazapine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Continue sertraline (Active Comparator): Continue sertraline at the dosage at 3 weeks
  Interventions: Drug: Sertraline
- Augment with mirtazapine (Active Comparator): Add mirtazapine to sertraline
  Interventions: Drug: Sertraline; Drug: Mirtazapine
- Switch to mirtazapine (Active Comparator): Stop sertraline and switch to mirtazapine
  Interventions: Drug: Mirtazapine

INTERVENTIONS:
Drug: Sertraline — Sertraline 50 mg/d or 100 mg/d for 6 more weeks
  Arms: Augment with mirtazapine; Continue sertraline
Drug: Mirtazapine — Augment with or switch to mirtazapine 15-45 mg/d
  Arms: Augment with mirtazapine; Switch to mirtazapine

SUMMARY:
The purpose of the study is to establish the optimum treatment strategy for first-line and second-line antidepressants in the acute phase treatment of major depression.

ELIGIBILITY:
Inclusion Criteria:

* non-psychotic unipolar major depressive episode (Diagnostic and Statistical Manual, Fourth Edition [DSM-IV]) in the preceding month
* age 25-75
* starting treatment with sertraline clinically indicated
* tolerability to sertraline 25 mg/d ascertained
* can understand and sign informed consent form
* can be contacted by telephone for symptom severity and adverse events

Exclusion Criteria:

* have received antidepressants, mood stabilizers, antipsychotics, psychostimulants, electroconvulsive therapy (ECT) or depression-specific psychotherapies in the preceding month
* history of schizophrenia, schizoaffective disorder or bipolar disorder
* current dementia, borderline personality disorder, eating disorder or substance dependence
* physical disease interfering with sertraline or mirtazapine treatment
* allergy to sertraline or mirtazapine
* terminal physical illness
* currently pregnant or breast-feeding
* high risk of imminent suicide
* requiring compulsory admission
* expected to change doctors within 6 months
* cohabiting relatives of research staff
* cannot understand Japanese

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2011 (Actual)
Dates: Start 2010-12; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Observer-rated depression severity (PHQ-9) | 9 weeks
  Personal Health Questionnaire-9 is a 9-item structured interview to measure depression severity. It will be rated by blinded telephone interview.

SECONDARY OUTCOMES:
Self-rated depression severity (BDI-II) | 9 weeks
  Beck Depression Inventory-II is a 21-item self-report of depression severity. It will be filled in by the patients themselves.
Global rating of side effects (FIBSER) | 9 weeks
  FIBSER stands for Frequency, Intensity and Burden of Side Effects Rating, which is an observer-rated global rating of side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Toshiaki A Furukawa, MD, PhD, Principal Investigator — Kyoto University Graduate School of Medicine / School of Public Health; Tatsuo Akechi, MD, PhD, Study Director — Nagoya City University Graduate School of Medical Sciences; Norio Watanabe, MD, PhD, Study Director — National Center of Neurology and Psychiatry, Japan; Shinji Shimodera, MD, PhD, Study Director — Kochi University Medical School; Mitsuhiko Yamada, MD, PhD, Study Director — National Center of Neurology and Psychiatry, Japan; Masatoshi Inagaki, MD, PhD, Study Director — Okayama University Graudate School of Medicine; Naohiro Yonemoto, MSc, Study Director — National Center of Neurology and Psychiatry, Japan; Kazuhira Miki, MD, PhD, Study Director — Miki Mental Clinic, Yokohama, Japan
Locations (2):
- Japan (2):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Kochi Medical School Hospital, Nangoku, Kochi

REFERENCES:
- [Derived] Kato T, Furukawa TA, Mantani A, Kurata K, Kubouchi H, Hirota S, Sato H, Sugishita K, Chino B, Itoh K, Ikeda Y, Shinagawa Y, Kondo M, Okamoto Y, Fujita H, Suga M, Yasumoto S, Tsujino N, Inoue T, Fujise N, Akechi T, Yamada M, Shimodera S, Watanabe N, Inagaki M, Miki K, Ogawa Y, Takeshima N, Hayasaka Y, Tajika A, Shinohara K, Yonemoto N, Tanaka S, Zhou Q, Guyatt GH; SUN☺D Investigators. Optimising first- and second-line treatment strategies for untreated major depressive disorder - the SUN☺D study: a pragmatic, multi-centre, assessor-blinded randomised controlled trial. BMC Med. 2018 Jul 11;16(1):103. doi: 10.1186/s12916-018-1096-5. PMID 29991347
- [Derived] Yonemoto N, Tanaka S, Furukawa TA, Kato T, Mantani A, Ogawa Y, Tajika A, Takeshima N, Hayasaka Y, Shinohara K, Miki K, Inagaki M, Shimodera S, Akechi T, Yamada M, Watanabe N, Guyatt GH; SUN(;_;)D Investigators. Strategic use of new generation antidepressants for depression: SUN(;_;) D protocol update and statistical analysis plan. Trials. 2015 Oct 14;16:459. doi: 10.1186/s13063-015-0985-6. PMID 26466684
- [Derived] Shimodera S, Kato T, Sato H, Miki K, Shinagawa Y, Kondo M, Fujita H, Morokuma I, Ikeda Y, Akechi T, Watanabe N, Yamada M, Inagaki M, Yonemoto N, Furukawa TA; SUN(;_;)D Investigators. The first 100 patients in the SUN(;_;)D trial (strategic use of new generation antidepressants for depression): examination of feasibility and adherence during the pilot phase. Trials. 2012 Jun 8;13:80. doi: 10.1186/1745-6215-13-80. PMID 22682213
- [Derived] Furukawa TA, Akechi T, Shimodera S, Yamada M, Miki K, Watanabe N, Inagaki M, Yonemoto N. Strategic use of new generation antidepressants for depression: SUN(;_;)D study protocol. Trials. 2011 May 11;12:116. doi: 10.1186/1745-6215-12-116. PMID 21569309